CLINICAL TRIAL: NCT03347045
Title: Trimodal Prehabilitation for Cystectomy Patients to Enhance Post-operative Care: A Randomized Control Trial
Brief Title: Trimodal Prehabilitation for Cystectomy Patients to Enhance Post-operative Care
Acronym: TPC-RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jason Martyn (Other)
Collaborators: Alberta Health services (Other); University of Calgary (Other); Physiotherapy Alberta - College + Association (Unknown); University of Alberta (Other)
Responsible Party: Sponsor-Investigator, Jason Martyn, Physiotherapist, Alberta Health Services, Calgary
Organization: Alberta Health Services, Calgary (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2017CRIF-JMARTYN
Record Dates: First submitted 2017-11-14; First posted 2017-11-20 (Actual); Last update posted 2017-11-20 (Actual); Status verified 2017-11

CONDITIONS: Bladder Cancer; Nutrition Aspect of Cancer
Keywords: cystectomy; nutrition; physiotherapy; prehabilitation; enhanced recovery after surgery
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — Single Person

STUDY DESIGN:
Intervention Model Description: Single-center pragmatic randomized-control trial.
Who Masked: Outcomes Assessor
Masking Description: Assessor blinding; due to the nature of the study, participant, care provider & investigator cannot be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Trimodal Prehab & ERP (Experimental): Trimodal prehab includes:
  1. Guided exercise program at Repsol Place in Calgary, Alberta 2x/week, hosted by the Total Cardiology group. Home-exercise program for another 3x/week.
  2. Nutritional optimization with a high-protein oral supplement, along with nutritional counseling and access to a Registered Dietitian on site.
  3. Anxiety reduction workshop and take-home anxiety reduction program.
  Interventions: Combination Product: Trimodal Prehab & ERP
- No Prehab; ERP Alone (Active Comparator): The active comparator group will be given a home exercise program, nutrition education, and a take-home anxiety reduction program.
  Interventions: Other: No Prehab; ERP Alone

INTERVENTIONS:
Combination Product: Trimodal Prehab & ERP — 1-hr daily exercise will be completed a total of 5d/week, of which 2 of these sessions are completed through a community fitness center. Following these sessions, the participant will consume a high-protein oral supplement.
  Additionally, during the program, participants will be given the option of attending a stress-reduction group and will receive a take-home anxiety-reduction program. They will have access to a physiotherapist, kinesiologist, registered dietitian, and physician throughout the program.
  The total length of this program is 8-weeks and is timed to occur in the waiting period between the consent for surgery and operation date.
  Other Names: Trimodal prehab and enhanced-recovery pathway (ERP) together
  Arms: Trimodal Prehab & ERP
Other: No Prehab; ERP Alone — 1-hr daily exercise with a self-completed home-exercise program. The participant will be given nutritional education material and a take-home anxiety-reduction program. They will be responsible for maintaining a journal of their activity.
  Other Names: No trimodal prehab; enhanced-recovery pathway (ERP) alone
  Arms: No Prehab; ERP Alone

SUMMARY:
Trimodal prehabilitation is a preoperative three-tiered (trimodal) approach to optimizing physical and mental health. It has been found to successfully improve functional recovery in patients undergoing colorectal surgery following an evidence-based enhanced-recovery pathway (ERP). It is unknown whether the same program is effective in patients undergoing a similar surgery for bladder cancer (radical cystectomy).

Objective: To evaluate the appropriateness of a standardized prehabilitation program for implementation into an enhanced recovery pathway for cystectomy patients and determine whether prehabilitation facilitates earlier recovery of functional capacity.

Hypothesis: Prehabilitation will ultimately improve recovery of functional capacity, clinical and patient-centered outcomes in patients undergoing radical cystectomy for bladder cancer.

Design: Participants will follow an 8-week trimodal prehabilitation program consisting of exercise therapy combined with nutritional counseling, protein supplementation, and psychological care; they will be compared to a cohort of participants following ERP care alone.

Conclusion: The proposal will provide insight into the feasibility and effectiveness of trimodal prehabilitation for radical cystectomy patients and may ultimately lead to improved clinical outcomes and reduced morbidity.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥ 18 years of age at time of consent for surgery.
2. Documentation of bladder cancer diagnosis as evidenced by diagnostic imaging and biopsy.
3. May or may not receive adjuvant therapy.
4. Written informed consent obtained from subject

Exclusion Criteria:

1. Presence of a condition or abnormality that in the opinion of the investigator would compromise the safety of the patient or adherence to the program. This includes:

   1. American Society of Anesthesiologists (ASA) health class status 4-5;
   2. Co-morbid medical, physical, and/or mental conditions including dementia, disabling orthopedic and neuromuscular disease, psychosis;
   3. Severe cardiac abnormalities, end-stage organ disease, sepsis, or morbid obesity (BMI greater than 35);
2. Undergoing radical cystectomy for a reason other than bladder cancer.
3. Poor comprehension of English or French
4. Screened by Total Cardiology staff and determined to be inappropriate for prehabilitation at their facility.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2018-01-15 (Estimated); Primary Completion 2019-01-15 (Estimated); Study Completion 2019-07-15 (Estimated)

PRIMARY OUTCOMES:
6-minute walk test (6MWT) | Multiple time-points over 20-weeks
  The 6MWT is a sub-maximal exercise test used to assess aerobic capacity and endurance. The distance covered over a time of 6 minutes is used as the outcome by which to compare changes in performance capacity.

SECONDARY OUTCOMES:
10-meter walk test (10mWT) | Multiple time-points over 20-weeks
  The 10 Metre Walk Test is a performance measure used to assess walking speed in metres per second over a short distance. It can be employed to determine functional mobility, gait, and vestibular function.
30s sit-to-stand test (30CST) | Multiple time-points over 20-weeks
  The 30CST is a measurement that assesses functional lower extremity strength in older adults. It is part of the Fullerton Functional Fitness Test Battery. This test was developed to overcome the floor effect of the 5 or 10 repetition sit to stand test in older adults.
Hand-grip dynamometry | Multiple time-points over 20-weeks
  A quantitative and objective measure of isometric muscular strength of the hand and forearm, predictive of overall upper-extremity function.
Functional Assessment of Cancer Therapy for Bladder Cancer (FACT-Bl)Questionnaire | Collected at beginning and end of 20-week participant involvement period
  A reliable and valid questionnaire that comprehensively assesses quality of life concerns pertinent to bladder cancer patients.
EuroQOL five dimensions (EQ-5D) Questionnaire | Collected at beginning and end of 20-week participant involvement period
  A short, generic quality of life questionnaire
Godin Leisure Time Exercise Questionnaire | Collected at beginning and end of 20-week participant involvement period
  A short questionnaire on self-reported physical activity.

OTHER OUTCOMES:
Length of hospital stay (LOS) | Collected at the finale of participant-involvement (20-weeks)
  Length of stay in the hospital starting from post-operative day #0 and terminating when the participant is discharged from the hospital.
30 day readmission rate | Collected at the finale of participant-involvement (20-weeks)
  Number of participants re-admitted to hospital within 30 days of discharge as a percentage of the total number of participants involved in the study.
Clavien-Dindo classification of Surgical Complications | Collected at the finale of participant-involvement (20-weeks)
  A classification scheme that objectively grades surgical complications using a descriptive grading system.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Martyn, MScPT, Principal Investigator — Alberta Health services

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (1):
  • Study Protocol (2017-11-11): https://cdn.clinicaltrials.gov/large-docs/45/NCT03347045/Prot_000.pdf